CLINICAL TRIAL: NCT05084209
Title: Preparing Patient-Caregiver Dyads with Parkinson's Disease for End-of-Life Decision Making
Brief Title: Preparing Patient-Caregiver Dyads with Parkinson's Disease for Future Decision Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Jiayun Xu, Assistant Professor, Purdue University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K23NR019099-01A1 (NIH)
Record Dates: First submitted 2021-09-25; First posted 2021-10-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
Keywords: end of life; medical decision making; advanced illness; family
MeSH Terms: conditions — Parkinson Disease; Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parkinson's medical decision making support intervention group (Experimental): All participants will complete an online medical decision making intervention, lasting about 60 minutes, and complete pre and post surveys.
  Interventions: Behavioral: Parkinson's medical decision making support

INTERVENTIONS:
Behavioral: Parkinson's medical decision making support — Participants will be asked to view and work through medical decision making support resources. The resources will include information on medical decisions that may occur in Parkinson's disease, and general medical decisions that anyone may need to make (i.e. choosing a medical decision maker). The resources will also include suggestions on how to discuss these decisions.

SUMMARY:
Persons with Parkinson's disease and family care partners are often unprepared to make difficult, future medical decisions. Earlier conversations about future medical decisions between persons with Parkinson's disease and family care partners are needed before communication and cognitive difficulties become severe. In this study, the investigators will pilot test a novel dyadic intervention to help persons with Parkinson's disease and family care partners make future medical decisions. The investigators hypothesize the intervention will be feasible and acceptable among persons with Parkinson's disease and family care partners.

DETAILED DESCRIPTION:
Investigators are looking for pairs of participants consisting of a person with a diagnosis of Parkinson's Disease, and a family care partner who is most likely to help make medical decisions in the future.

For this study, pairs will complete a survey to understand how engaged participants are in discussing future medical decisions, demographics, and the severity of Parkinson's disease. This survey will take about 15 minutes. Then, participants will work through a medical decision making support intervention together. Completing the intervention in-person, on the phone, or via video conferencing is acceptable. The resources will provide information on future medical decisions participants may need to make. The intervention is completely online and will take about 60 minutes to complete. Participants will have 2 weeks to complete the intervention.

The investigators will call participants a week after enrollment to ask about technical difficulties completing the intervention, provide assistance with intervention material navigation as needed, and answer questions about the intervention. Participants will receive another online survey 2 weeks after enrollment to understand engagement in discussing future medical decisions, and acceptability of the intervention. The 2 week survey will take about 15 minutes to complete.

ELIGIBILITY:
Person with Parkinson's Disease Inclusion Criteria:

* Self-report a clinical diagnosis of Parkinson Disease
* Does not have a diagnosis of dementia
* Speak and read English
* Have access to a reliable phone or internet connection
* Have access to an online connection through a smartphone, tablet, or computer device
* Be comfortable navigating websites or have someone available to assist
* Agree to be audio recorded during intervention

Care Partner Inclusion Criteria:

* Self-identify as the family member who will likely make medical decisions for the person with Parkinson Disease in the future OR who is the legally appointed health care representative
* Self-report not having a diagnosis of dementia
* Speak and read English
* Have access to a reliable phone or internet connection
* Have access to an online connection through a smartphone, tablet, or computer device
* Be comfortable navigating websites or have someone available to assist
* Agree to be audio recorded during intervention

Exclusion Criteria:

* Cannot see well enough to see words on a newspaper even with corrective lenses
* Used the intervention resources before
* If cognition is questionable and cannot pass consent understanding questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline Advance Care Planning Engagement Survey at 2 weeks | Baseline, 2 weeks post intervention
  Assesses knowledge, contemplation, self-efficacy, and readiness on a 5-point Likert scale.
Intervention feasibility/acceptability | 2 weeks post intervention
  Ratings of ease of use, helpfulness, and likeliness of recommending the intervention to others on Likert-scales.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayun Xu, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No